CLINICAL TRIAL: NCT00320047
Title: Effects of Baclofen on Binge Eating in Bulimia Nervosa and Binge Eating Disorder
Brief Title: Effectiveness of Baclofen in the Treatment of People With Bulimia Nervosa or Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #5017; R21MH065024 (NIH); DNBBS 72-NBR
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-09

CONDITIONS: Eating Disorders; Bulimia Nervosa
Keywords: Binge Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participants will take baclofen for 10 weeks.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Participants will take baclofen 3 times a day, before meals, for 10 weeks. Baclofen dosages will be low to begin, followed by a gradual increase over a 2-week period. Upon reaching the maximum tolerated dose of baclofen, participants will continue at this dosage level until Week 11, at which time the dose will be gradually decreased. If any serious side effects occur, baclofen dosage will be decreased to the previous tolerated dosage level.

SUMMARY:
This study will evaluate the effectiveness of the drug baclofen in reducing binge eating and associated food cravings in people with bulimia nervosa or binge eating disorder.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) and binge eating disorder (BED) are serious eating disorders that are characterized by frequent uncontrolled eating binges. Binge eating is associated with both psychological and physical health problems, such as depression, obesity, stomach problems, and heart problems. Treatment options for binge eating, however, are limited. Baclofen, a drug that enhances the GABA-B neurotransmitter's ability to inhibit neuronal activity in the brain, is commonly used as a muscle relaxant. It has also been shown, however, to have positive effects on binge eating when used in animals and on substance abuse when used in humans. This study will evaluate the effectiveness of baclofen in reducing binge eating and associated food cravings in people with BN or BED.

People interested in participating in this study will first report to the study site for two initial visits, which will involve blood tests and interviews regarding medical history. If eligible, participants will take part in this 13-week open-label study. Participants will take baclofen 3 times a day, before meals, for 10 weeks. Baclofen dosages will be low to begin, followed by a gradual increase over a 2-week period. Upon reaching the maximum tolerated dose of baclofen, participants will continue at this dosage level until Week 11, at which time the dose will be gradually decreased. If any serious side effects occur, baclofen dosage will be decreased to the previous tolerated dosage level. Participants will also keep a daily record of any episodes of binge eating. Study visits will be held biweekly. At each visit, participants will be interviewed by a psychiatrist about their mental health history and eating patterns, and will fill out questionnaires about their eating habits, emotional states, and any side effects. Phone interviews will be conducted during the weeks in between study visits.

ELIGIBILITY:
Inclusion Criteria:

For people with BN:

* Meets DSM-IV criteria for BN
* Disease duration is more than 1 year
* Self-induces vomiting
* Weighs between 80 and 120% of ideal weight
* Binge eats on at least 6 days during the 2-week run-in period

For obese people with BED:

* Meets DSM-IV criteria for BED
* Obese (body mass index [BMI] is greater than 30 kg/m²)
* Binge eats on at least 6 days during the 2-week run-in period

Exclusion Criteria:

For all participants:

* Significant medical illness
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder as defined by DSM-IV-TR
* Moderate to severe depression as defined by a score greater than 18 on the Hamilton Depression Scales
* Current DSM-IV-TR diagnosis of organic mental disorder, factitious disorder, or malingering
* History of a personality disorder (e.g., schizotypal, borderline, or antisocial) that might interfere with assessment or compliance with the study procedures
* At risk for suicide
* Currently taking medication other than birth control pills or over-the-counter medication
* History of drug or alcohol abuse within 3 months prior to study entry
* Pregnant, planning to become pregnant, or breast feeding
* Known intolerance to baclofen, or related muscle relaxants
* Orthostatic hypotension

Additional exclusion criteria for people with BN:

* Underweight (BMI less than 18 kg/m²)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Frequency of binge eating | Measured at Week 13

SECONDARY OUTCOMES:
Cravings associated with binge eating | Measured at Week 13

CONTACTS AND LOCATIONS:
Overall Officials: B. T. Walsh, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (1):
- Eating Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States